CLINICAL TRIAL: NCT04605900
Title: Impact of Therapeutic Footwear and Plantar Orthoses for Patients With Diabetic Neuropathic Foot in Quality of Life and Functionality: A Interventional Study
Brief Title: Impact of Therapeutic Footwear and Plantar Orthoses on Diabetic Neuropathic Foot in Quality of Life and Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Algarve (Other)
Collaborators: University of Huelva (Other); OKM Química Ortopédica S.L. (Unknown); Lola - J. Andrade Ferreira Neves Lda (Unknown); Instituto São João de Deus (ISJD) (Unknown); Ortobalance - Ortopedia Técnica e Desportiva (Unknown); Sensor Médica (Unknown); Pierre Fabre Portugal (Unknown); Associação para o Estudo da Diabetes Mellitus e de Apoio ao Diabético do Algarve (AEDMADA) (Unknown); Unidade Funcional de Faro - Agrupamento de Centros de Saúde do Central (Unknown)
Responsible Party: Principal Investigator, Marta Botelho, Research Fellowship, Universidade do Algarve
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0348_CIE_6_E
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Peripheral Neuropathy
Keywords: Quality of life; Postural Balance; Functionality; Foot Orthoses; Footwear
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A pre and post-test analysis was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Footwear (SF) (Experimental): Intervention: plantar orthoses, education on foot self-care and appropriate standard footwear.
  Interventions: Device: Standard Footwear; Device: Plantar Orthoses; Behavioral: Education on foot self-care
- Orthopedic Footwear (OF) (Experimental): Intervention: plantar orthoses, education on foot self-care and orthopedic footwear.
  Interventions: Device: Orthopedic Footwear; Device: Plantar Orthoses; Behavioral: Education on foot self-care

INTERVENTIONS:
Device: Orthopedic Footwear — The orthopedic footwear used by the OF Group was manufactured by the company J. Andrade Ferreira Neves Lda. with materials suitable for the diabetic foot, as registered with INFARMED under registration ID 279515.
  Arms: Orthopedic Footwear (OF)
Device: Standard Footwear — In the SF Group, it was recommended to use standard shoes more suitable for diabetic foot, with some specific characteristics, such as sports or walking shoes. The acquisition or not of a more suitable shoes by the participants was at the discretion of each individual.
  Arms: Standard Footwear (SF)
Device: Plantar Orthoses — The plantar orthoses (PO) that both groups used for distribute of plantar loads was based on the principle of total contact. The confection material consisted in a liner of EVA shore 20º and polyurethane filling ELAX flexible (expandable) from OKM Química Ortopédica SL.
Behavioral: Education on foot self-care — An information leaflet with foot care was delivered, with the aim of ensuring that participants were informed about the care they should continually take with their feet during the study period. This leaflet was created based on the guidelines of the "Associação Protetora dos Diabéticos" in Portugal.

SUMMARY:
This study determines the effectiveness of plantar orthoses and custom-made orthopedic footwear in functional level and quality of life of persons with diabetes type 2 and diabetic peripheral neuropathy. This study is important due the loss of protective sensation, feet are vulnerable to minor trauma caused by plantar pressure as well as mechanical and thermal injuries. Thus, Plantar Orthoses become necessary to reduce PP and align the foot. Additionally, it is known that footwear is the most frequent cause of diabetic foot injury, since ulceration is frequently a consequence of the continuous trauma provoked by inadequate footwear. For a higher efficacy in the treatment of the foot, it is also necessary to use custom-made orthopedic footwear, indicated in the treatment of foot pathologies.

The lack of studies that evaluate the impact of this treatment on clinical measures such as quality of life and functional level, led to the development of this study, comparing a standard treatment (standard footwear and plantar orthoses) with an optimal treatment suggested in diabetic foot guidelines (therapeutic footwear and plantar orthoses).

DETAILED DESCRIPTION:
This clinical trial includes 2 parallel intervention groups with a pre- and post-test analysis. In the standard footwear (SF) group, plantar orthoses, standard footwear and education on foot self-care were applied and in the orthopedic footwear (OF) group the same intervention was applied, but with orthopedic footwear.

Both intervention groups were evaluated at two different time points, with the pre-test taking place at the beginning of the study (T0 - Baseline) and the post-test taking place 4 months after the application of the treatment (T4). In the middle of the study, at two months (T2) a questionnaire was applied in order to understand the adherence and the perception of individuals about the intervention applied.

The screening of diabetic peripheral neuropathy was made with the Michigan Neuropathy Screening Instrument (MNSI) and the description of the sample with an evaluation questionnaire.

The FL was evaluated through the Lower Extremity Functional Scale (LEFS), physical tests and the postural, static and dynamic barometric assessment. QoL was assessed with SF-36 and the adherence and satisfaction with a questionnaire created ad hoc.

ELIGIBILITY:
Inclusion Criteria:

* Presence of type 2 DM;
* Have at least 6 months from diagnosis of DM;
* Presence of Diabetic Polyneuropathy;
* No history of plantar orthoses and orthopedic footwear use.

Exclusion Criteria:

* Active ulceration;
* Severe osteoarticular deformities;
* Presence of cognitive impairment;
* Gait with technical devices;
* Diagnosis of neurological pathology that can affect the gait pattern;
* Diagnosis of another pathology that can negatively influence the study: depression, the presence of uncontrolled cardiovascular diseases and active cancer.
* Surgical interventions on the spine and lower limbs, with less than 1 year of recovery.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Change the Quality of Life | 4 months
  Significantly change any subscore or total score of Medical Outcomes Study 36-item Short-Form Health Survey instrument, that was use it to assess quality of life. Instrument scores can range between 0 - 100. Higher values mean better self-perception of quality of life.
Change the Performance of Lower Extremity Functional Scale | 4 months
  Change at least 9 points in Lower Extremity Functional Scale (minimum change for clinically relevant functional improvement). Instrument scores can range between 0 - 80. Higher values mean better functionality.
Change the Functional Reach Test performance | 4 months
  Significantly change the maximum distance (cm) attained in Functional Reach Test.
Change the Unipedal Stance Test performance | 4 months
  Change the time (s) in left and right unipedal stance.
Change the Static Full Tandem Test performance | 4 months
  Change the time (s) in full-tandem position.
Change the Walking Full Tandem Test performance | 4 months
  Achieve at least 10 steps in full-tandem.
Change the Time Up and Go Test performance | 4 months
  Change the time (s) in performing the Time Up and Go test.
Change the 6 minutes walk test performance | 4 months
  Change the distance (m) covered for 6 minutes of walking.

SECONDARY OUTCOMES:
Change the Postural Stability (length displacement of Center of Pressure) | 4 months
  Significantly change the length displacement (mm) of center of pressure.
Change the Postural Stability (displacement of Center of Pressure) | 4 months
  Significantly change the amplitude mediolateral and anteroposterior displacement (mm) of Center of Pressure.
Change the Postural Stability (Ellipse surface) | 4 months
  Significantly change the ellipse surface (mm2).
Change the Postural Stability (Mean Speed of Center of Pressure) | 4 months
  Significantly change the mean speed of CoP (mm/s).
Change the Postural Stability (Standard deviation of Center of Pressure) | 4 months
  Significantly change the mediolateral and anteroposterior standard deviation (mm).
Change the Postural Stability (Root Mean Square) | 4 months
  Significantly change the root mean square index (mm).
Change the Postural Stability (Romberg Ration Index) | 4 months
  Significantly change the romberg ration index (mm).
Change the mean pressure in static position | 4 months
  Change the mean pressure (kPa) on each foot in static position.
Change the maximum pressure in static position | 4 months
  Change the maximum pressure (kPa) in each forefoot and hindfoot in static position.
Change the support surface in static position | 4 months
  Change the support surface (cm2) between the plantar surface and the platform sensors, during the support phase on each of the feet.
Change the load distribution in static position | 4 months
  Change the load distribution (%) between each foot.
Change the maximum pressure in gait | 4 months
  Change the maximum pressure (kPa) of each foot in gait.
Change the mean pressure in gait | 4 months
  Change the mean pressure (kPa) on each foot in gait.
Change the plantar impression length in gait | 4 months
  Change the plantar impression Length (mm) of each of the feet.
Change the support surface in gait | 4 months
  Change the support surface (cm2) of each foot.
Change the longitude of CoP in gait | 4 months
  Change the longitude of the center of pressure (mm) of each foot.
Change the load distribution in gait | 4 months
  Change the load distribution (%) between the forefoot and hindfoot and between the medial and lateral zone.
Change the foot progression angle of gait | 4 months
  Change the foot progression angle in gait.
Change the double support time of gait | 4 months
  Change the double support time (ms) in gait.
Change the support time of gait | 4 months
  Change the support time (ms) for each foot in gait.
Change the step length of gait | 4 months
  Change the step length (m) in gait.
Adherence to the intervention | 2 months
  Number of hours per day using the devices (telephone monitoring).
Self-Perception of improvements | 2 months
  Presence or not of improvements in feet/legs with the devices (telephone monitoring).
Satisfaction with devices | 2 months
  Level of Satisfaction (totally satisfied, quite satisfied, satisfied, little satisfied, dissatisfied) with the devices (telephone monitoring).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Botelho, PhD, Principal Investigator — Researcher
Locations (1):
- Marta Botelho, Faro, Algarve, Portugal